CLINICAL TRIAL: NCT06049134
Title: Immunogenicity and Clinical Efficacy of 20-valent Pneumococcal Conjugate Vaccine (PCV20) in Lymphoma Survivors After Treatment With Anti-CD20 Therapy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-0590; NCI-2023-07264 (Other: NCI-CTRP Clinical Trials Gov)
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm Group A (PCV20) (Experimental): Participants will receive 1 dose of the vaccine
  Interventions: Biological: PCV20
- Arm Group B (PCV20) (Experimental): Participants will receive 2 doses of the vaccine
  Interventions: Biological: PCV20

INTERVENTIONS:
Biological: PCV20 — Given by Injection into the muscle

SUMMARY:
To compare the effects of a pneumococcal vaccine called PCV20 when given as a single dose versus a boosted regimen to patients who previously received anti-CD20 therapy as treatment for B cell lymphoma.

DETAILED DESCRIPTION:
Primary Objectives:

--Compare the humoral responses in terms of difference in IgG titers at 1 month from routine single dose PCV20 or a boosted PCV20 regimen in B cell lymphoma survivors who previously received treatment with anti-CD20 therapy.

Secondary Objectives:

* Compare the humoral responses in terms of difference in IgG titers at 3, 6 and12 from routine single dose PCV20 or a boosted PCV20 regimen in B cell lymphoma survivors who previously received treatment with anti-CD20 therapy.
* Estimate the rate of pneumonia (all bacterial pneumonia including pneumococcal pneumonia) within a year from routine single dose PCV20 or a boosted PCV20 regimen in lymphoma survivors who previously received treatment with anti-CD 20 therapy.
* Correlate humoral responses to development of bacterial pneumonia and pneumococcal pneumonia and with severity of this infection in lymphoma survivors within a year of vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have a history of non-Hodgkin B-cell lymphoma and whose disease has been in remission for at least 1 year.
2. Patients who received any anti-CD20 therapy at any time during their treatment for B-cell lymphoma.
3. Patients who are at least 18 years of age.
4. Patients who can provide consent; no legal authorized representative will be able to provide consent on a patient's behalf.

Exclusion Criteria:

1. Patients who have received cellular therapy, including chimeric antigen receptor T-cell therapy or any type of hematopoietic cell transplantation.
2. Patients who have received PCV or pneumococcal polysaccharide vaccine within 5 years of screening for enrollment.
3. Patients who are unable to attend follow-up appointments at designated times at MD Anderson.
4. Any vulnerable population patient ((children, pregnant women, cognitively impaired adults, or prisoners)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Fareed Khawaja, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org